CLINICAL TRIAL: NCT00955656
Title: Delta Primary Care Provider (PCP) Survey on Asthma Management
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 110132
Record Dates: First submitted 2009-08-06; First posted 2009-08-10 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Asthma
Keywords: Characteristics of medical practices; Practitioners providing care to children with asthma; Medically underserved and impoverished Arkansas Delta region; Characteristics of medical practices and practitioners; Disadvantaged populations
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- primary care providers: Primary care providers who receive the survey will be the primary care provider identified by study participants enrolled in our ongoing study entitled, "Asthma in the Delta Region of Arkansas: Characterization of Disease and Impact of Environmental Factors" (ARIA#53054)

SUMMARY:
The proposed study will utilize a survey format to examine the attitudes, perceptions, and practices of primary care providers in the Delta region of Arkansas.

DETAILED DESCRIPTION:
Study Design. Primary care providers will be sent a providers packet to include a cover letter explaining the survey and its purpose as well as a 2-part questionnaire that includes nine selected short patient vignettes and a questionnaire regarding their personal and practice characteristics.

Study Population. Individuals who receive the survey will be the primary care provider identified by study participants enrolled in our ongoing study entitled, "Asthma in the Delta Region of Arkansas: Characterization of Disease and Impact of Environmental Factors" (ARIA#53054). We will send the survey to all identified practitioners in Lee, Phillips, Desha, Chicot, St. Francis, and surrounding counties. Future studies will include primary care providers from other Arkansas Delta counties pending funding.

Inclusion/Exclusion Criteria. We will send the survey to all identified practitioners in Lee, Phillips, Desha, Chicot, St. Francis, and surrounding counties. Future studies will include primary care providers from other Arkansas Delta counties pending funding.

Instruments. Delta Primary Care Provider Survey. The self administered survey examines the attitudes, perceptions and practices of primary care providers. The 2-part questionnaire includes nine selected short patient vignettes and a questionnaire regarding the providers personal and practice characteristics.

ELIGIBILITY:
Inclusion Criteria:

* We will send the survey to all identified practitioners in Lee, Phillips, Desha, Chicot, St. Francis, and surrounding counties.
* Future studies will include primary care providers from other Arkansas Delta counties pending funding.

Exclusion Criteria:

* None.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who receive the survey will be the primary care provider identified by study participants enrolled in our ongoing study entitled, "Asthma in the Delta Region of Arkansas: Characterization of Disease and Impact of Environmental Factors" (ARIA#53054).
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The proposed study will utilize a survey format to examine the attitudes, perceptions, and practices of primary care providers in the Delta region of Arkansas. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tamara T. Perry, M.D., Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Hospital Research Institute, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.